CLINICAL TRIAL: NCT05561283
Title: Evaluation of the Satisfaction and Relevance of Leadership Training for Residents - START Study
Brief Title: Evaluation of the Satisfaction and Relevance of Leadership Training for Residents
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1273
Record Dates: First submitted 2022-09-21; First posted 2022-09-30 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life; Medical Residents
Keywords: leadership; meditation; residents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of residents (Experimental): Medical residents undergoing the leadership and meditation training
  Interventions: Diagnostic Test: Self-questionnaires

INTERVENTIONS:
Diagnostic Test: Self-questionnaires — Self-questionnaires on satisfaction, burn-out, depression, anxiety, relational skills and sleep quality

SUMMARY:
Health students are the future actors of the health system. They are exposed to many stressors in their journey. The quality of life of medical students is alarming worldwide: 11.1% of undergraduate and postgraduate residents reportedly have suicidal ideation and 27.2% have depressive symptoms. In addition, 44.2% suffer from burn-out syndrome. In the third cycle, 28.8% suffer from depressive symptoms and 35.1% from burn-out syndrome. This finding is shared internationally among medical residents. Health professionals are facing a global problem which it is crucial to act.

At national level, a survey on the mental health of young doctors carried out in 2017 found, among the 7603 residents who responded a prevalence: 22.8% of depressive symptoms, 59.7% of anxiety symptoms, 23.4% of suicidal thoughts, including 5.0% in the month prior to the survey. In 2018, a French report on the quality of life of health by Dr Donata Marra highlighted a real malaise affecting residents and the need to intervene "for residents, for carers and for patients", through the implementation of specific recommendations. The proposal 6 of the report emphasises the prevention of psychosocial risks through educational interventions such as training in collaborative management. On a personal level, the aim is to the leadership of each individual, in terms of stress management, communication, cross-disciplinary skills or even the introduction of relational simulations in the teaching of an awareness of deviant behaviour and harassment. The stress factors are indeed multiple during health studies confrontation with death, competition, increasing responsibilities… Perceived stress has a negative impact on the quality of life and burnout. Effective stress management strategies could therefore help to improve the quality of life of residents.

In this context, the analysis of the literature highlights three main areas of intervention that could contribute to resident leadership in favour of their quality of life: stress management, healthy living and the construction of a professional identity.

The Junior Leadership programme for residents from the beginning of their professional formation designed to provide basic knowledge and skills in healthcare leadership and to develop cross-disciplinary skills. The aim is to provide the necessary support for the success of the resident's professional project by participating in the improvement of their quality of life and the prevention of psycho-social risks.

The study therefore propose to evaluate the feasibility of training in leadership and meditation on the satisfaction of resident.

ELIGIBILITY:
Inclusion Criteria:

* residents assigned to the Hospices Civils de Lyon
* Informed consent given by the resident

Exclusion Criteria:

* Pregnant women, women in labour or nursing mothers
* Persons deprived of their liberty by a judicial or administrative decision
* Persons under psychiatric care
* Persons of full age who are subject to a legal protection measure (guardianship, curatorship)
* Persons who are not affiliated to a social security scheme or who are beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Description of the satisfaction on the Junior Leadership programme for residents evaluated by the questionnaire recommanded by the HAS | At 4 months (at the end of the training that lasts around 4 months)
  The satisfaction of the residents will be evaluated by a self-questionnaire according to model recommended by the Haute Autorité de Santé (HAS)and used in the framework of the SAMSEI programme (SAMSEI="Stratégies d'Apprentissage des Métiers de Santé en Environnement Immersif" that means in English "Learning Strategies for Healthcare Professions in an Immersive Environment") and the Lyon South Health Simulation Centre. The questionnaire will evaluate the interest, practical usefulness, density of information information, conformity with the objectives, the material conditions of the training, the activity of the participants and the motivation to continue the training.

SECONDARY OUTCOMES:
Change of proportion of burn-out evaluated the Maslach's burn-out inventory scale | Before training (baseline) and 3 months, 6 months and 1 year after training
  The proportion of residents showing symptoms of burn-out will be assessed by the Maslach's burn-out inventory before training and 3 months, 6 months and 1 year after training.
Change int he presence of symptoms of anxiety and depression evaluated by the HADS scale | Before training (baseline) and 3 months, 6 months and 1 year after training
  Anxiety and depression symptoms will be assessed by Hospital Anxiety and Depression Scale (HADS) before training and at 3 months, 6 months and 1 year after training.
Change of the real-life stress levels in the professional environment of residents evaluated by the Karasek scale | Before training (baseline) and 3 months, 6 months and 1 year after training
  The stress of residents in their work environment will be assessed using the Karasek scale, which evaluates psychosocial risk factors at work before training and at 3 months, 6 months and and 1 year after the training
Change of relational skills evaluated by Cungi and Rey's communication scale | Before training (baseline) and 3 months, 6 months and 1 year after training
  Caregivers' interpersonal skills will be assessed by Cungi and Rey's communication scale at 3 months, 6 months and 1 year after the training.
Change of sleep quality of the residents evaluated by the LEEDS scale | Before training (baseline) and 3 months, 6 months and 1 year after training
  The sleep quality of the residents will be assessed by the LEEDS scale before training and at 3 months, 6 months and 1 year after training
Change of the use of psychoactive substances by residents collected by questionnaire | Before training (baseline) and 3 months, 6 months and 1 year after training
  The use of psychoactive substances will be collected from residents before the training and at 3 months, 6 months and 1 year after the training
Change of the use of medical/psychological by residents collected by questionnaire | Before training (baseline) and 3 months, 6 months and 1 year after training
  The use of medical/psychological support will be collected from residents before the training and at 3 months, 6 months and 1 year after the training.
Change of the number of days off for sikness collected by questionnaire | Before training (baseline) and 3 months, 6 months and 1 year after training
  The number of days off sick will be collected from the residents before the training and at 3 months, 6 months and 1 year after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle de simulation en Santé de Lyon Sud (PL3S), Oullins, France

IPD SHARING:
Plan to Share IPD: No